CLINICAL TRIAL: NCT01576393
Title: Adolescent Involvement in Parental Substance Abuse Treatment: Evaluation of EBFT
Brief Title: Adolescent Involvement in Parental Substance Abuse Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Natasha Slesnick, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006B0269; R01DA023062 (NIH)
Record Dates: First submitted 2012-04-09; First posted 2012-04-12 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Substance Abuse
Keywords: substance abuse; treatment; families
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Home-Based family therapy (Experimental): 12 home-based family therapy sessions
  Interventions: Behavioral: Home-based Family Therapy
- Office-based family therapy (Active Comparator): 12 office-based family therapy sessions
  Interventions: Behavioral: office-based family therapy
- Women's Health Education (Placebo Comparator): 12 womens's health education sessions
  Interventions: Behavioral: WHE

INTERVENTIONS:
Behavioral: Home-based Family Therapy — 12 home-based family therapy sessions
  Other Names: home-based Ecologically-based Family therapy
  Arms: Home-Based family therapy
Behavioral: office-based family therapy — 12 office-based family therapy sessions
  Other Names: Office-based Ecologically-based Family Therapy
  Arms: Office-based family therapy
Behavioral: WHE — 12 Women's Health Education Sessions
  Other Names: Women's Health Education Intervention
  Arms: Women's Health Education

SUMMARY:
Given the reciprocal nature of parent-child interaction, involvement of the adolescent in their mother's substance abuse treatment plan might be associated with reductions in adult relapse and improvements in child functioning. These findings would support the assertion that focus on family dynamics in substance abuse treatment programs is an effective use of resources and an important target of intervention efforts. One hundred eighty-three substance abusing mothers and their child (n=61 assigned to each condition) will receive treatment as usual (TAU) and be randomly assigned to 1) Ecologically-based family therapy (EBFT) conducted in the home or 2) Ecologically-based family therapy conducted at the treatment center, or 3) an attention control, Women's Health Education (WHE). In order to examine the endurance of treatment effects, this project will assess the parent and child at 3, 6, 12, and 18 months post-baseline.

Hypotheses

1. It is expected that 1) mothers and children assigned to home and office based family therapy will show greater reductions in substance use and improvement in individual and family functioning at post-treatment compared to those in the attention control, and 2) those assigned to home-based family therapy will show greater reductions in substance use and improved individual and family functioning at post-treatment compared to those assigned to office-based family therapy.
2. It is expected that 1) those assigned to home or office based family therapy will continue to maintain improvements in substance use, individual and family domains over time (time by treatment interaction) compared to those assigned to the attention control and 2) those assigned to home-based family therapy will continue to maintain improvements in substance use, individual and family domains over time (time by treatment interaction) compared to those assigned to office-based family therapy.
3. It is hypothesized that improved family interaction skills will mediate substance use, individual and family outcomes.
4. It is expected that EBFT in the home and EBFT in the office will be more cost effective than TAU, and that EBFT in the home will be more cost effective than EBFT in the office

DETAILED DESCRIPTION:
Many researchers have studied the effects of parental alcohol and drug use on child outcomes. These studies conclude that parental substance use has the potential to negatively impact children's psychosocial development by depriving them of adequate care and supervision, impeding their socioemotional and cognitive development and/or influencing them to become substance users as well. Considering a bidirectional, systemic model for understanding the development, maintenance and recovery of substance use problems, it follows that the child impacts parents' behaviors as well. Family therapy has consistently shown that involvement of family members in the treatment of substance users is associated with higher levels of engagement and retention in treatment. Many studies report pre to post treatment reductions in substance use and related problems among those receiving couples and family therapy. While randomized clinical trials of family therapy have involved adult identified patients (IPs) in couples therapy and adolescent IPs in family therapy, this study will evaluate a family systems intervention involving an 8-16 year old child in the treatment plan of the adult treatment seeker. In the current study, alcohol and drug treatment seeking adult mothers of a child (8-16) living in the home will be engaged. All clients will be randomized to (1) ecologically-based family therapy (EBFT) in the home + treatment as usual (TAU), (2) EBFT at the office + TAU, or (3) TAU + attention control. The relative efficacy of this approach will be evaluated at 3, 6, 12, and 18 months post-baseline. Proposed change mechanisms (mediators) for family therapy will be evaluated. Differential treatment response as a function of gender, family history of alcohol or drug use, and primary alcohol v. drug abuse (moderators) will be investigated to better understand the intervention. The study will also examine how, if at all, treatment engagement and retention impact parent and adolescent response to treatment. Information gained through this project will help evaluate the utility of including adolescent family members in the treatment plan of their adult parents. Finally, the study will include an economic evaluation component to estimate the economic cost of each intervention and determine which condition is most cost effective. Intervention that includes a focus on parent-child interaction has the potential to enhance substance use reductions, reduce parent relapse, and improve family and emotional health among adults. Involvement of the child offers the opportunity to increase the potential protection of a positive parent-child relationship which is shown to be associated with positive developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult mothers seeking outpatient treatment for alcohol or drug abuse or dependence as measured using the computerized diagnostic interview schedule (CDIS; Shaffer, 1992), and who report substance use within the past 90 days
2. A child, between the ages of 8 to 16, lives with the mother at least 50% time over the prior 2 years or continuously for the 6 months prior to the assessment interview.
3. If more than one 8-16 year old lives in the home, the one with the greater problem severity will be included in the study. Substance use will be probed ("Have you ever used alcohol or drugs?"). If one youth answers yes, and the other answers no, the one who answers yes will be included. If both child answer "yes", then the Form 90 substance use section [history and current pattern] will be administered to each. The child who reports the more severe pattern and history of use [age of onset, type of drug used, frequency of current use] will be included. If neither youth reports using alcohol or drugs, then the Youth Self-Report (Achenbach & Edelbrock, 1982) will be administered and the youth with the greater total problem score will be included.
4. Family lives within 60 miles of the treatment facility.
5. Child and adult agree to participate in the assessment and treatment intervention.

Exclusion Criteria:

1. Evidence of unremitted psychosis or other condition which would impair their ability to understand and participate in the intervention or consent for research participation (as determined by CDISC).

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2009-08; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Substance use | baseline, 3, 6, 12 and 18-months
  Change in frequency of reported substance use

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Slesnick, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States